CLINICAL TRIAL: NCT04606953
Title: Working Memory Training With Attention Process Training (APT-II) in Older Adults With Mild Cognitive Impairment : Impacts on Cognition and Ecological Activities
Brief Title: Working Memory Training in Older Adults With Mild Cognitive Impairment : Impacts on Cognition and Ecological Activities
Acronym: APT-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Paris 5 - Rene Descartes (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Sophie Blanchet, Ph D, Director of these and Associate professor, University of Paris 5 - Rene Descartes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APT-II Project
Record Dates: First submitted 2020-07-16; First posted 2020-10-28 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
Keywords: mild cognitive impairment; Alzheimer's disease; memory impairment; working memory training; cognitive rehabilitation; Aging
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Memory Disorders

STUDY DESIGN:
Intervention Model Description: In this single-blind, randomized controlled trial, patients are randomly assigned to either a "cognitive training" experimental group (n=15) or a "standard care" control group (n=15).
Who Masked: Outcomes Assessor
Masking Description: In this single-blind, randomized controlled trial, the follow-up action evaluator is in a blind condition. The evaluator does not know the group to which the participants belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Process Training (APT-II) (Experimental): Patients in the experimental group receive the APT-II training program (Attention Process Training) individually with a psychologist for 8 weeks (2 sessions/week). The exercises target different attentional components and working memory in the auditory-visual modalities. They are of increasing difficulty while being adapted to each patient's profile in order to maximize the effects on cognitive reserve. During the sessions, the emphasis is on generalizing the gains towards the most problematic daily activities in order to reduce the impact of the patients' cognitive problems in their daily lives.
  Interventions: Behavioral: Attention Process Training (APT-II)
- Standard care (No Intervention): Patients in the control group receive standard routine care.

INTERVENTIONS:
Behavioral: Attention Process Training (APT-II) — The exercises target different attentional components and working memory in the auditory-visual modalities. They are of increasing difficulty while being adapted to the profile of each patient in order to maximize the effects on cognitive reserve. During the sessions, the emphasis is on generalizing the gains to the most problematic daily activities in order to reduce the impact of cognitive disorders in patients' daily life.
  Arms: Attention Process Training (APT-II)

SUMMARY:
Older adults with Mild Cognitive Impairment (MCI) have an increased risk of developing dementia but do not meet the criteria for dementia. Cognitive rehabilitation makes it possible to compensate, at least in part, for cognitive deficits with the ultimate goal of reducing their impact in everyday life. The objective of the research is to evaluate the short- and long-term effectiveness and generalization of an attention and working memory training program (APT-II) on cognition and ecological activities in MCI patients with a randomized controlled trial. Thirty MCI patients will be randomly assigned between a "cognitive training with APT-II" condition and a control (routine care) condition. The intervention will consist of an 8-week individual cognitive training program (2 sessions/week), training different attentional components and working memory. This has the advantage of insisting on the transfer of the acquired knowledge in sessions to daily activities. To evaluate the effectiveness of the treatment, cognitive and functional follow-up measures (including a virtual reality task) are administered at several time intervals. This project should contribute to better management of cognitive disorders by offering a new standardized rehabilitation tool in French to clinical practice.

DETAILED DESCRIPTION:
Older adults with Mild Cognitive Impairment (MCI) have an increased risk of developing dementia, but do not meet the criteria for dementia. Some of these individuals nevertheless remain in a stable state or even return to the norm. Currently, pharmacological treatments have not been shown to be sufficiently effective in treating cognitive deficits. The major challenge is to identify other therapeutic approaches to reduce the risk of cognitive impairment progressing to dementia. Deficits in working memory, which are very common in these individuals, have a prognostic value for progression to dementia of the Alzheimer's type. Cognitive re-education makes it possible to compensate, at least in part, for cognitive disorders with the ultimate goal of reducing their repercussions in daily life. Executive control training can improve working memory and attention, but how this gain is transferred to activities of daily living (ADLs) remains poorly understood to date. The generalization of cognitive gains to ADLs is crucial, however, as this generalization may contribute to patients' functional autonomy.

This project aims to evaluate the effectiveness of attention and working memory training (APT-II) on cognitive function and ecological activities in MCI patients by means of a single-blind randomized controlled trial. Working memory is involved in information manipulation and attentional processes. This ability is called upon in higher cognitive functions such as language, reasoning, comprehension, but also in various complex ADL situations. Deficits in working memory thus contribute significantly to other cognitive or functional impairments in MCI patients. To date, some working memory training has been shown to have an immediate impact on working memory in this population. However, long-term maintenance and impact on daily life have not been demonstrated in this population. Researchers of this study propose to fill this gap by using the APT-II (or Attention Process Training) program, which focuses on the transfer of cognitive gains from the start of training. Indeed, the APT-II program was translated from English to French by the scientific coordinator (S. Blanchet). The English version has already been validated in various populations with mild cognitive dysfunction following brain injury, stroke or small vessel brain disease. The efficacy of APT-II has never been studied in older adults with IBD. For the first time a research team evaluate the short- and long-term efficacy of this program in MCI patients on cognition and ADLs using virtual reality. This new technology provides an ecological and objective measure for the evaluation of memory and other cognitive functions while simulating naturalistic and controlled situations. The objective is therefore to evaluate the effectiveness of an attention and working memory training program (APT-II) on cognitive function in patients with MCI. To achieve this objective, patients with MCI are randomly assigned to an APT-II program or to a control group. Cognitive training with the APT-II program will include progressively more difficult and adaptive exercises and will be varied to facilitate near and far cognitive transfer. Attention, working memory and episodic memory are measured at different time intervals (before, immediately after, 3 and 6 months after training). A unique feature of the cognitive training program is its emphasis on generalization by teaching participants how to maximize the transfer of the attention management strategies learned during the sessions to their various ADLs requiring attention and executive control. Homework exercises targeting these different cognitive functions in ADLs are also provided between sessions.

The protocol is offered to elderly people with mild cognitive impairment. In this single-blind randomized controlled trial, participants are randomly assigned either to a "cognitive training" experimental group (n=20) or a "standard care" control group (n=20). Recruitment is multi-centric, and takes place via memory consultations from several sites: Tenon Hospital (collaboration with Dr Eric Bouvard), AP-HP Sorbonne University, and Dr Mettling's private neurology practice (Paris XI). MCI patients are selected according to the criteria of Petersen (2004). A battery of standardized neuropsychological tests is first administered to ensure that participants meet our criteria. Patients must be at least 55 years of age and have an impairment of attention, exécutive, memory and/or working memory as evidenced by impaired performance on tests assessing attention or executive function (score 1.5 standard deviation below the norm on these tests). Participants meeting the selection criteria are invited to continue the study. The project has already been approved by the Committee for the Protection of Persons (CPP) EST-III of the ANSM (BCR ID: 2018-A02377-48, N°CPP: 18.11.05, N° 18.08.21.66617). Patients in the experimental group receive the APT-II training program individually with a psychologist for 8 weeks (2 sessions/week). The exercises target different attentional components and working memory in the auditory-visual modalities. This exercices are of increasing difficulty while being adapted to each patient's profile in order to maximize the effects on cognitive reserve. During the sessions, the emphasis is on generalizing the gains towards the most problematic daily activities in order to reduce the impact of the patients' cognitive problems in their daily lives. Patients in the control group receive standard routine care. In order to test the impact of the APT-II training program on cognitive function and daily activities, cognitive and functional follow-up measures are administered in a blind condition just before (T0), after (T1), and 3 (T2) and 6 months (T3) after the intervention. The last two measures will be used to study long-term maintenance of earnings. The cognitive follow-up measures will test the effects of near (attention, working memory) and far (episodic memory) cognitive transfers and generalization to daily activities with questionnaires. Functional follow-up measures include a virtual reality task assessing episodic memory in the presence of interferences in order to examine the effects of training on an ecological situation with high demands on attentional resources.

MCI patients who received the APT-II training program should perform better on attention and working memory tasks after training, with a distant transfer to episodic memory tasks compared to the control group who received standard care during the training time interval. Following cognitive training, MCI patients should also be less susceptible to environmental interferences as assessed with the virtual reality task, while reporting fewer cognitive complaints in everyday life with maintenance of these gains over time. In patients in the control group, it is anticipated that there will be no difference in follow-up measures between the different times or the presence of decreased performance as these patients are at risk of developing neurodegenerative pathology. In a preliminary study evaluating the efficacy of the APT-II programme by the same team of research, six MCI patients (m = 68 ± 10.56 years) attended 10 sessions of the APT-II programme (2 sessions/week). Statistical analyses indicate that after cognitive training, MCI patients tended to improve their performance on a working memory task (upside down number span, p = .06). There was also a gain in daily activities and well-being, as assessed by the Cognitive Failure Questionnaire (p = .04) and the Bravo Wellness Questionnaire (p = .04), respectively. These encouraging results support the effectiveness of the APT-II program in IBD patients. They remain to be confirmed on larger samples with a randomized controlled trial. This project could provide the clinic with a standardized cognitive intervention tool for better cognitive management of these patients. The clinical impact of the project will hopefully be significant.

ELIGIBILITY:
Inclusion Criteria:

* MCI criteria according to Petersen 2004
* 55 years and over
* Native French-speaking or bilingual participant living in the Paris region
* Normal or corrected vision and hearing
* Presence of episodic memory and/or attention and/or working memory impairment as evidenced by substandard performance on neuropsychological test(s) evaluating these processes (-1.5 deviations from the norms)

Exclusion Criteria:

* Presence of dementia
* Significant impact of cognitive impairment on activities of daily living requiring external assistance or institutionalization
* Stroke or brain injury
* Presence of moderate to severe psychiatric disorders
* Ethylism
* General anesthesia in the last six months
* Treatment directly impacting cognition
* Patient with significant depression (cut off GDS > 10)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Mini Mental State MMSE | Prior the program
  The mini-mental state (MMS) or mini-mental state examination (MMSE) or Folstein test is a test for the evaluation of global cognitive functions. This test is used for diagnostic purposes when there is a suspicion of dementia and cognitive disorders. It evaluates temporospatial orientation, memory, attention, language and praxies. Folstein, Folstein and McHugh, 1975; Greco version.
Mini Mental State MMSE | Immediately after the program
  The mini-mental state (MMS) or mini-mental state examination (MMSE) or Folstein test is a test for the evaluation of global cognitive functions. This test is used for diagnostic purposes when there is a suspicion of dementia and cognitive disorders. It evaluates temporospatial orientation, memory, attention, language and praxies. Folstein, Folstein and McHugh, 1975; Greco version.
Mini Mental State MMSE | 3 months follow-up
  The mini-mental state (MMS) or mini-mental state examination (MMSE) or Folstein test is a test for the evaluation of global cognitive functions. This test is used for diagnostic purposes when there is a suspicion of dementia and cognitive disorders. It evaluates temporospatial orientation, memory, attention, language and praxies. Folstein, Folstein and McHugh, 1975; Greco version.
Mini Mental State MMSE | 6 months follow-up
  The mini-mental state (MMS) or mini-mental state examination (MMSE) or Folstein test is a test for the evaluation of global cognitive functions. This test is used for diagnostic purposes when there is a suspicion of dementia and cognitive disorders. It evaluates temporospatial orientation, memory, attention, language and praxies. Folstein, Folstein and McHugh, 1975; Greco version.
Digit span | Prior the program
  The Digit span task is a test evaluating the phonological loop and executive control capabilities of the working memory. The test consists of hearing a series of numbers orally by the examiner and must repeat the same series in the same order or in reverse. This test measures the limited capabilities of a specialized verbal short-term memory system described by Baddeley and Hitch (1974). WAIS-III Weschler,2000 and MEM-III Weschler 2001
Digit span | Immediately after the program
  The Digit span task is a test evaluating the phonological loop and executive control capabilities of the working memory. The test consists of hearing a series of numbers orally by the examiner and must repeat the same series in the same order or in reverse. This test measures the limited capabilities of a specialized verbal short-term memory system described by Baddeley and Hitch (1974). WAIS-III Weschler,2000 and MEM-III Weschler 2001
Digit span | 3 months follow-up
  The Digit span task is a test evaluating the phonological loop and executive control capabilities of the working memory. The test consists of hearing a series of numbers orally by the examiner and must repeat the same series in the same order or in reverse. This test measures the limited capabilities of a specialized verbal short-term memory system described by Baddeley and Hitch (1974). WAIS-III Weschler,2000 and MEM-III Weschler 2001
Digit span | 6 months follow-up
  The Digit span task is a test evaluating the phonological loop and executive control capabilities of the working memory. The test consists of hearing a series of numbers orally by the examiner and must repeat the same series in the same order or in reverse. This test measures the limited capabilities of a specialized verbal short-term memory system described by Baddeley and Hitch (1974). WAIS-III Weschler,2000 and MEM-III Weschler 2001
PASAT (Naegele and Mazza, 2004) | Prior the program
  PASAT is a test that evaluates information processing skills, sustained attention, and shared attention. The individual hears numbers in succession with an interval of 4 seconds. He must add the last digit heard to the last given without losing his attention.
PASAT (Naegele and Mazza, 2004) | Immediately after the program
  PASAT is a test that evaluates information processing skills, sustained attention, and shared attention. The individual hears numbers in succession with an interval of 4 seconds. He must add the last digit heard to the last given without losing his attention.
PASAT (Naegele and Mazza, 2004) | 3 months follow-up
  PASAT is a test that evaluates information processing skills, sustained attention, and shared attention. The individual hears numbers in succession with an interval of 4 seconds. He must add the last digit heard to the last given without losing his attention.
PASAT (Naegele and Mazza, 2004) | 6 months follow-up
  PASAT is a test that evaluates information processing skills, sustained attention, and shared attention. The individual hears numbers in succession with an interval of 4 seconds. He must add the last digit heard to the last given without losing his attention.
Brown Peterson's Paradigm (Peterson and Peterson, 1959) | Prior the program
  Experimental technique to study forgetting in short-term memory and also used as a measure of the central administrator of working memory. The task is to present the subjects with sequences of three consonants. After the presentation of each sequence, the subject is asked to either perform an immediate recall of the consonants or to perform a countdown task from 30 seconds, 20 seconds or 10 seconds. At the end of this count, the subject must give the series again starting from 3 consonants.
Brown Peterson's Paradigm (Peterson and Peterson, 1959) | Immediately after the program
  Experimental technique to study forgetting in short-term memory and also used as a measure of the central administrator of working memory. The task is to present the subjects with sequences of three consonants. After the presentation of each sequence, the subject is asked to either perform an immediate recall of the consonants or to perform a countdown task from 30 seconds, 20 seconds or 10 seconds. At the end of this count, the subject must give the series again starting from 3 consonants.
Brown Peterson's Paradigm (Peterson and Peterson, 1959) | 3 months follow-up
  Experimental technique to study forgetting in short-term memory and also used as a measure of the central administrator of working memory. The task is to present the subjects with sequences of three consonants. After the presentation of each sequence, the subject is asked to either perform an immediate recall of the consonants or to perform a countdown task from 30 seconds, 20 seconds or 10 seconds. At the end of this count, the subject must give the series again starting from 3 consonants.
Brown Peterson's Paradigm (Peterson and Peterson, 1959) | 6 months follow-up
  Experimental technique to study forgetting in short-term memory and also used as a measure of the central administrator of working memory. The task is to present the subjects with sequences of three consonants. After the presentation of each sequence, the subject is asked to either perform an immediate recall of the consonants or to perform a countdown task from 30 seconds, 20 seconds or 10 seconds. At the end of this count, the subject must give the series again starting from 3 consonants.
Virtual reality memory task | Prior the program
  A developed virtual reality task was also administered to the participants to allow a more ecological analysis of episodic memory and divided attention.
Virtual reality memory task | Immediately after the program
  A developed virtual reality task was also administered to the participants to allow a more ecological analysis of episodic memory and divided attention.
Continious Performance task CPT | Prior the program
  CPT is a task of sustained and selective attention on the computer. The task consists of clicking on the space bar of the computer when a letter is presented on the screen except for the letter "X". The person should not click if they see the letter "X" presented. This test takes several minutes.
Continious Performance task CPT | Immediately after the program
  CPT is a task of sustained and selective attention on the computer. The task consists of clicking on the space bar of the computer when a letter is presented on the screen except for the letter "X". The person should not click if they see the letter "X" presented. This test takes several minutes.

SECONDARY OUTCOMES:
Cognitive Failure Questionnaire | Prior the program
  The Cognitive Failure Questionnaire (CFQ) is a questionnaire that evaluates daily cognitive failures.
Cognitive Failure Questionnaire | Immediately after the program
  The Cognitive Failure Questionnaire (CFQ) is a questionnaire that evaluates daily cognitive failures.
Cognitive Failure Questionnaire | 3 months follow-up
  The Cognitive Failure Questionnaire (CFQ) is a questionnaire that evaluates daily cognitive failures.
Cognitive Failure Questionnaire | 6 months follow-up
  The Cognitive Failure Questionnaire (CFQ) is a questionnaire that evaluates daily cognitive failures.
Bravo's Scale | Prior the program
  This scale is a measure of general well-being. The questionnaire contains 18 items that determine how the respondent feels. The first fourteen questions are answered on a 6-point Likert scale (0-5) and the last four questions on a 10-point scale (0-10) to give a maximum score of 110.
  A high well-being score is close to 110.
Bravo's Scale | Immediately after the program
  This scale is a measure of general well-being. The questionnaire contains 18 items that determine how the respondent feels. The first fourteen questions are answered on a 6-point Likert scale (0-5) and the last four questions on a 10-point scale (0-10) to give a maximum score of 110.
  A high well-being score is close to 110.
Bravo's Scale | 3 months follow-up
  This scale is a measure of general well-being. The questionnaire contains 18 items that determine how the respondent feels. The first fourteen questions are answered on a 6-point Likert scale (0-5) and the last four questions on a 10-point scale (0-10) to give a maximum score of 110.
  A high well-being score is close to 110.
Bravo's Scale | 6 months follow-up
  This scale is a measure of general well-being. The questionnaire contains 18 items that determine how the respondent feels. The first fourteen questions are answered on a 6-point Likert scale (0-5) and the last four questions on a 10-point scale (0-10) to give a maximum score of 110.
  A high well-being score is close to 110.
APT-II Attention Questionnaire | Prior the program
  The attention questionnaire is a questionnaire of the attention complaint felt by the subject in everyday life. This questionnaire is taken from the APT program.
APT-II Attention Questionnaire | Immediately after the program
  The attention questionnaire is a questionnaire of the attention complaint felt by the subject in everyday life. This questionnaire is taken from the APT program.
APT-II Attention Questionnaire | 3 months follow-up
  The attention questionnaire is a questionnaire of the attention complaint felt by the subject in everyday life. This questionnaire is taken from the APT program.
APT-II Attention Questionnaire | 6 months follow-up
  The attention questionnaire is a questionnaire of the attention complaint felt by the subject in everyday life. This questionnaire is taken from the APT program.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie SB Blanchet, Ph.D, Study Director — University of Paris
Locations (1):
- SABA, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baddeley A, Logie R, Bressi S, Della Sala S, Spinnler H. Dementia and working memory. Q J Exp Psychol A. 1986 Nov;38(4):603-18. doi: 10.1080/14640748608401616. No abstract available. PMID 3809575
- [Background] Barker-Collo SL, Feigin VL, Lawes CM, Parag V, Senior H, Rodgers A. Reducing attention deficits after stroke using attention process training: a randomized controlled trial. Stroke. 2009 Oct;40(10):3293-8. doi: 10.1161/STROKEAHA.109.558239. Epub 2009 Jul 23. PMID 19628801
- [Background] Belleville S, Boller B. Comprendre le stade compensatoire de la maladie d'Alzheimer et agir pour promouvoir la cognition et la plasticite cerebrale. Can J Exp Psychol. 2016 Dec;70(4):288-294. doi: 10.1037/cep0000087. PMID 27936842
- [Background] Blanchet S, McCormick L, Belleville S, Gely-Nargeot MC, Joanette Y. [Mild cognitive impairments in the elderly: a critical review]. Rev Neurol (Paris). 2002 Jan;158(1):29-39. French. PMID 11938320
- [Background] Kim H, Chey J, Lee S. Effects of multicomponent training of cognitive control on cognitive function and brain activation in older adults. Neurosci Res. 2017 Nov;124:8-15. doi: 10.1016/j.neures.2017.05.004. Epub 2017 Jun 1. PMID 28577979
- [Background] Palmese CA, Raskin SA. The rehabilitation of attention in individuals with mild traumatic brain injury, using the APT-II programme. Brain Inj. 2000 Jun;14(6):535-48. doi: 10.1080/026990500120448. PMID 10887887
- [Background] Petersen RC, Smith GE, Waring SC, Ivnik RJ, Tangalos EG, Kokmen E. Mild cognitive impairment: clinical characterization and outcome. Arch Neurol. 1999 Mar;56(3):303-8. doi: 10.1001/archneur.56.3.303. PMID 10190820
- [Background] Petersen RC, Lopez O, Armstrong MJ, Getchius TSD, Ganguli M, Gloss D, Gronseth GS, Marson D, Pringsheim T, Day GS, Sager M, Stevens J, Rae-Grant A. Author response: Practice guideline update summary: Mild cognitive impairment: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology. Neurology. 2018 Aug 21;91(8):373-374. doi: 10.1212/WNL.0000000000006042. No abstract available. PMID 30126885
- [Background] Plancher G, Gyselinck V, Piolino P. The Integration of Realistic Episodic Memories Relies on Different Working Memory Processes: Evidence from Virtual Navigation. Front Psychol. 2018 Jan 30;9:47. doi: 10.3389/fpsyg.2018.00047. eCollection 2018. PMID 29441037
- [Background] Saba M, Blanchet S. [Working memory training in normal and pathological aging: neurocognitive gains and generalization]. Geriatr Psychol Neuropsychiatr Vieil. 2020 Jun 1;18(2):187-195. doi: 10.1684/pnv.2020.0860. French. PMID 32554350
- [Background] Simon SS, Tusch ES, Feng NC, Hakansson K, Mohammed AH, Daffner KR. Is Computerized Working Memory Training Effective in Healthy Older Adults? Evidence from a Multi-Site, Randomized Controlled Trial. J Alzheimers Dis. 2018;65(3):931-949. doi: 10.3233/JAD-180455. PMID 30103334
- [Background] Telonio A, Blanchet S, Maganaris CN, Baltzopoulos V, Villeneuve S, McFadyen BJ. The division of visual attention affects the transition point from level walking to stair descent in healthy, active older adults. Exp Gerontol. 2014 Feb;50:26-33. doi: 10.1016/j.exger.2013.11.007. Epub 2013 Nov 27. PMID 24291246
- [Background] Murray LL, Keeton RJ, Karcher L. Treating attention in mild aphasia: evaluation of attention process training-II. J Commun Disord. 2006 Jan-Feb;39(1):37-61. doi: 10.1016/j.jcomdis.2005.06.001. Epub 2005 Jul 21. PMID 16039661
- [Background] Unsworth N, Fukuda K, Awh E, Vogel EK. Working memory and fluid intelligence: capacity, attention control, and secondary memory retrieval. Cogn Psychol. 2014 Jun;71:1-26. doi: 10.1016/j.cogpsych.2014.01.003. Epub 2014 Feb 14. PMID 24531497